CLINICAL TRIAL: NCT05055674
Title: Randomized Controlled Trial Testing the Effects of Motherly: a Standalone Smartphone Application Treatment for Women With Postpartum Depression
Brief Title: The Effects of Motherly on Postpartum Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Guilherme Vanoni Polanczyk, MD PhD, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OR2019-62903
Record Dates: First submitted 2021-08-31; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Postpartum Depression
Keywords: postpartum depression; smartphone application; digital technology; maternal depression; mental health; mental disorder
MeSH Terms: conditions — Depression, Postpartum; Psychological Well-Being; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two groups: a) intervention, which will have access to the Motherly app; or b) active control, which will be given access to COMVC, a smartphone app that delivers only psychoeducational content.
Who Masked: Outcomes Assessor
Masking Description: Participants will be aware of the intervention received, as well as investigators and professionals responsible for monitoring app usage during the study. The Outcome assessor will be blind to randomization status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motherly App (Experimental): Participants in this arm will have access to Motherly, a smartphone app that is designed to promote life habits that have been shown to improve depression and mental health in mothers.
  Interventions: Behavioral: Motherly app
- COMVC App (Active Comparator): Participants in this arm will have access to COMVC, a smartphone app designed to deliver only psychoeducational content and mental health monitoring.
  Interventions: Behavioral: COMVC app

INTERVENTIONS:
Behavioral: Motherly app — The Motherly app is organized in four different modules: 1) Library: a collection of brief texts on several topics related to health and pregnancy, 2) Health: journeys with varying degrees of interactivity designed to teach and engage participants in well-established psychological techniques (behavioral activation, cognitive restructuring, emotion regulation, stress management techniques, mindfulness and meditation, sleep hygiene techniques), 3) Pregnancy and motherhood: a module to help mothers keep track of their health care visits, medical exams, and their childrens' development, and 4) Profile: a module allowing participants to keep track of activities and goals completed in the Health module journeys, and to assess depression and anxiety symptoms with brief questionnaires, with results displayed graphically in a timeline and in the the form of short feedback texts.
  Arms: Motherly App
Behavioral: COMVC app — The COMVC displays over 30 brief psychoeducational videos on several topics related to general mental health, such as depression, anxiety, stress, sleep, problem solving techniques, among others. Psychoeducation is limited to video only (no interactivity). The content of these videos was developed by clinicians, researchers, and professors from the Psychiatry Department of the Medical School of the University of Sao Paulo and from the Federal University of Rio Grande do Sul. Mental health monitoring is delivered by means of brief questionnaires assessing depression and anxiety symptoms, which can be filled at users' discretion. Users' responses are displayed graphically in a timeline and they receive short feedback texts based on assessment results.
  Arms: COMVC App

SUMMARY:
Investigators will be test the efficacy of Motherly, a smartphone application (app) to treat depression in women with postpartum Depression. The Motherly app offers psychoeducation, mood and anxiety monitoring, several well-established psychological techniques (behavioral activation, cognitive restructuring, emotion regulation, stress management techniques, mindfulness and meditation, sleep hygiene), and helps mothers organize their medical appointments and keep track of their childrens' development. The efficacy of the Motherly app will be tested in a parallel two-arm randomized controlled trial. Participants will be randomly allocated to receive the Motherly app (intervention), or COMVC (active control), a smartphone app that delivers only psychoeducational content related to general mental health.

DETAILED DESCRIPTION:
The postpartum period is strongly associated with increased risk for depression, with estimates of approximately 19% of women affected by the disorder. Psychosocial interventions such as home visiting programs and well-established psychological therapies are efficient to treat this condition but require a significant number of qualified trained professionals. However, financial and human resources to meet these demands are scarce in developing countries such as Brazil. Therefore, interventions delivered via electronic devices such as smartphones might fill this gap. Our objective is to test the efficacy of Motherly, a smartphone application (app) to treat depression in women with postpartum Depression. The Motherly app offers psychoeducation, mood and anxiety monitoring, several well-established psychological techniques (behavioral activation, cognitive restructuring, emotion regulation, stress management techniques, mindfulness and meditation, sleep hygiene), and helps mothers organize their medical appointments and keep track of their childrens' development. The efficacy of the Motherly app will be tested in a parallel two-arm randomized controlled trial. Two-hundred and sixty-four (N=264) 18-40-years-old women with postpartum depression will be to one of two groups: (1) intervention, which will have access to the Motherly app; or (2) active control, which will be given access to COMVC, a smartphone app that delivers only psychoeducational content on general mental health (COMVC means "With You" in Brazilian Portuguese). Duration of treatment will be four weeks, during which participants in both groups will be assessed at the beginning (baseline; T0), end (post treatment, T1), and 1 month after treatment completion (follow-up, T2).

ELIGIBILITY:
Inclusion Criteria:

* Women who had given birth to a live baby in the past 12 months;
* Age between 18-40 years;
* Edinburgh Postnatal Depression Scale (EPDS) total score ≥ 10;
* Depression symptoms present in the past 2 weeks;
* Being literate;
* Owing an Android or iPhone smartphone for personal use.

Exclusion Criteria:

* Intellectual, visual, or auditory deficiency;
* Chronic diseases that prevent using smartphones or understanding how to use the apps;
* Severe and/or chronic mental health diagnosis (schizophrenia or bipolar disorder).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 264 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms | Posttreatment (T1) 1 month after baseline
  Change in mean total scores between intervention and control groups in the Edinburgh Postnatal Depression Scale (EPDS) at Posttreatment (T1)

SECONDARY OUTCOMES:
Depression symptoms | Follow-up (T2) 2 months after baseline
  Change in mean total scores between intervention and control groups in the Edinburgh Postnatal Depression Scale (EPDS)
Anxiety symptoms | Posttreatment (T1) 1 month after baseline and Follow-up (T2) 2 months after baseline
  Change in mean total scores between intervention and control groups in the General Anxiety Disorder-7 (GAD-7)
Sleep quality | Posttreatment (T1) 1 month after baseline and Follow-up (T2) 2 months after baseline
  Change in mean total scores between intervention and control groups in the Single-item Sleep Quality Scale at Posttreatment (T1) and Follow-up (T2).
Quality of Life: Physical Health | Posttreatment (T1) 1 month after baseline and Follow-up (T2) 2 months after baseline
  Change in "Physical Health Quality of Life" mean scores between intervention and control groups in the 12-item health survey (SF-12) at Posttreatment (T1) and Follow-up (T2).
Quality of Life: Mental Health | Posttreatment (T1) 1 month after baseline and Follow-up (T2) 2 months after baseline
  Change in "Mental Health Quality of Life" mean scores between intervention and control groups in the 12-item health survey (SF-12) at Posttreatment (T1) and Follow-up (T2).
Parenting stress | Posttreatment (T1) 1 month after baseline and Follow-up (T2) 2 months after baseline
  Change in "Total Stress" mean scores between intervention and control groups in the Parenting Stress Index (PSI) Short Form at Posttreatment (T1) and Follow-up (T2).
Parental Distress | Posttreatment (T1) 1 month after baseline and Follow-up (T2) 2 months after baseline
  Change in "Parental Distress" mean scores between intervention and control groups in the Parenting Stress Index (PSI) Short Form at Posttreatment (T1) and Follow-up (T2).
Parent-child Dysfunctional Interaction | Posttreatment (T1) 1 month after baseline and Follow-up (T2) 2 months after baseline
  Change in "Parent-child Dysfunctional Interaction" mean scores between intervention and control groups in the Parenting Stress Index (PSI) Short Form at Posttreatment (T1) and Follow-up (T2).
Difficult Child | Posttreatment (T1) 1 month after baseline and Follow-up (T2) 2 months after baseline
  Change in "Difficult Child" mean scores between intervention and control groups in the Parenting Stress Index (PSI) Short Form at Posttreatment (T1) and Follow-up (T2).
Attachment | Posttreatment (T1) 1 month after baseline and Follow-up (T2) 2 months after baseline
  Change in "Attachment" mean scores between intervention and control groups in the Parenting Stress Index (PSI) Short Form at Posttreatment (T1) and Follow-up (T2).
Parenting Competence | Posttreatment (T1) 1 month after baseline and Follow-up (T2) 2 months after baseline
  Change in "Competence" mean scores between intervention and control groups in the Parenting Stress Index (PSI) Short Form at Posttreatment (T1) and Follow-up (T2).

OTHER OUTCOMES:
Activation and avoidance behaviors | Posttreatment (T1) 1 month after baseline and Follow-up (T2) 2 months after baseline
  Change in mean scores between intervention and control groups in the The Behavioral Activation for Depression Scale-Short Form (BADS-SF) scale.
Reinforcement probability and environmental suppression | Posttreatment (T1) 1 month after baseline and Follow-up (T2) 2 months after baseline
  Change in mean scores between intervention and control groups in the Reward Probability Index (RPI) scale.
Response to treatment | Posttreatment (T1) 1 month after baseline and Follow-up (T2) 2 months after baseline
  Comparison between intervention and control groups according to two categories: Very much improved, Much improved, Minimally improved vs. No change, Minimally worse, Much worse, Very much worse, in the Clinical Global Impression Index (CGI) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme V Polanczyk, MD, PhD, Principal Investigator — Professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gelaye B, Rondon MB, Araya R, Williams MA. Epidemiology of maternal depression, risk factors, and child outcomes in low-income and middle-income countries. Lancet Psychiatry. 2016 Oct;3(10):973-982. doi: 10.1016/S2215-0366(16)30284-X. Epub 2016 Sep 17. PMID 27650773
- [Background] Wang L, Wu T, Anderson JL, Florence JE. Prevalence and risk factors of maternal depression during the first three years of child rearing. J Womens Health (Larchmt). 2011 May;20(5):711-8. doi: 10.1089/jwh.2010.2232. Epub 2011 Mar 22. PMID 21426237
- [Background] Jacques N, Mesenburg MA, Matijasevich A, Domingues MR, Bertoldi AD, Stein A, Silveira MF. Trajectories of maternal depressive symptoms from the antenatal period to 24-months postnatal follow-up: findings from the 2015 Pelotas birth cohort. BMC Psychiatry. 2020 May 14;20(1):233. doi: 10.1186/s12888-020-02533-z. PMID 32408866
- [Background] Matijasevich A, Murray J, Cooper PJ, Anselmi L, Barros AJ, Barros FC, Santos IS. Trajectories of maternal depression and offspring psychopathology at 6 years: 2004 Pelotas cohort study. J Affect Disord. 2015 Mar 15;174:424-31. doi: 10.1016/j.jad.2014.12.012. Epub 2014 Dec 13. PMID 25553403
- [Background] Zuccolo PF, Xavier MO, Matijasevich A, Polanczyk G, Fatori D. A smartphone-assisted brief online cognitive-behavioral intervention for pregnant women with depression: a study protocol of a randomized controlled trial. Trials. 2021 Mar 23;22(1):227. doi: 10.1186/s13063-021-05179-8. PMID 33757591
- [Background] Weisel KK, Fuhrmann LM, Berking M, Baumeister H, Cuijpers P, Ebert DD. Standalone smartphone apps for mental health-a systematic review and meta-analysis. NPJ Digit Med. 2019 Dec 2;2:118. doi: 10.1038/s41746-019-0188-8. eCollection 2019. PMID 31815193
- [Background] Santos IS, Matijasevich A, Tavares BF, Barros AJ, Botelho IP, Lapolli C, Magalhaes PV, Barbosa AP, Barros FC. Validation of the Edinburgh Postnatal Depression Scale (EPDS) in a sample of mothers from the 2004 Pelotas Birth Cohort Study. Cad Saude Publica. 2007 Nov;23(11):2577-88. doi: 10.1590/s0102-311x2007001100005. PMID 17952250
- [Background] Goncalves H, Pearson RM, Horta BL, Gonzalez-Chica DA, Castilho E, Damiani M, Lima RC, Gigante DP, Barros FC, Stein A, Victora CG. Maternal depression and anxiety predicts the pattern of offspring symptoms during their transition to adulthood. Psychol Med. 2016 Jan;46(2):415-24. doi: 10.1017/S0033291715001956. Epub 2015 Oct 12. PMID 26456404
- [Background] Netsi E, Pearson RM, Murray L, Cooper P, Craske MG, Stein A. Association of Persistent and Severe Postnatal Depression With Child Outcomes. JAMA Psychiatry. 2018 Mar 1;75(3):247-253. doi: 10.1001/jamapsychiatry.2017.4363. PMID 29387878
- [Background] Kingston D, Tough S, Whitfield H. Prenatal and postpartum maternal psychological distress and infant development: a systematic review. Child Psychiatry Hum Dev. 2012 Oct;43(5):683-714. doi: 10.1007/s10578-012-0291-4. PMID 22407278
- [Background] Grote NK, Bridge JA, Gavin AR, Melville JL, Iyengar S, Katon WJ. A meta-analysis of depression during pregnancy and the risk of preterm birth, low birth weight, and intrauterine growth restriction. Arch Gen Psychiatry. 2010 Oct;67(10):1012-24. doi: 10.1001/archgenpsychiatry.2010.111. PMID 20921117